CLINICAL TRIAL: NCT03117062
Title: Evaluation of Postoperative Pain Intensity Following Occlusal Reduction in Teeth Associated With Symptomatic Irreversible Pulpitis and Symptomatic Apical Periodontitis: A Randomized Clinical Study
Brief Title: Occlusal Reduction and Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Radwa Sameeh Emara, assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEBC-CU-2015-15-166
Record Dates: First submitted 2017-04-06; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occlusal Reduction (Experimental): performing occlusal reduction on functional cusps until abscence of contact was confirmed
  Interventions: Other: occlusal reduction
- non-occlusal reduction (No Intervention): occlusal surface left intact

INTERVENTIONS:
Other: occlusal reduction — relief of occlusion following endodontic treatment
  Other Names: occlusal relief
  Arms: Occlusal Reduction

SUMMARY:
The purpose of this randomized clinical study was to evaluate the impact of occlusal reduction on the incidences of post-instrumentation and post-obturation pain. Forty four patients were included in this study. Inclusion criteria were posterior mandibular teeth having symptomatic irreversible pulpitis and symptomatic apical periodontitis. Patients were randomized into two equal groups. In the intervention group the functional and nonfunctional cusps were reduced until absence of contact was confirmed, while in the control group the occlusal surfaces were left intact. Standard endodontic treatment was performed in two visits using rotary nickel titanium files for shaping, 2.5% sodium hypochlorite for cleaning and lateral condensation technique with resin sealer for obturation. Pain was assessed preoperatively, then after 6, 12, 24 and 48 hours following instrumentation, then after 6 and 12 hours following obturation. Visual Analogue Scale (VAS) was used as the primary outcome measure. Patients were given a placebo to be administrated in case of severe pain and ibuprofen 400mg was prescribed in case of persistent pain.

DETAILED DESCRIPTION:
Recruitment of the study participants was done from the outpatient clinic of the Endodontic Department of the Faculty of Oral and Dental Medicine, Cairo University.

Randomization was done to assign participants to the study groups by chance and not choice. 44 numbers were generated and randomly allocated to either intervention or control group on a table using Microsoft Office Excel 2010. Each participant was given a number from 1 to 44 according to his turn in enrollment in the study.

Root canal treatment was completed in two visits. Before treatment, each patient was given pain scale chart and was asked to record their pain level. The tooth was anesthetized using inferior alveolar nerve block technique by local anesthesia of 1.8 - 3.6 ml of 2% Mepivacaine HCl. The access cavity preparation was performed using round carbide bur and Endo-z bur. After access cavity in the intervention group, all occlusal contacts on the functional and non-functional cusps as well as on the marginal ridges were reduced using a wheel diamond bur. Absence of contact was confirmed using an articulating paper. In the control group, all occlusal contacts were left intact. The tooth was then properly isolated with rubber dam. The patency of the root canals was confirmed using stainless steel hand K-files size #10 and #15. Working length was determined using an electronic apex locator and confirmed radiographically to be 1 mm shorter than radiographic apex. Mechanical preparation was done by crown-down technique using rotary Revo-S instruments and Ethylene Diamine Tetra Aceticacid gel as a lubricant. The canals were thoroughly irrigated using 3ml of 2.5% sodium hypochlorite following each instrument. After dryness of the canals using paper points, a cotton pellet was placed in the pulp chamber and the access cavity was sealed with a temporary filling. After 7 days, the root canals were obturated with lateral condensation technique using 0.04 taper gutta-percha and AdSeal resin-based root canal sealer.

Degree of postoperative pain was measured using visual analogue scale (VAS) after 6, 12, 24 and 48 hours after instrumentation then at 6 and 12 hours after obturation. The VAS consists of a 10-cm line anchored by two extremes "No pain" and "pain as bad as could be". The patients were asked to choose the mark that represents their level of pain. Pain level was assigned to one of four categorical scores: 1, None(0); 2,Mild(1-3); 3,Moderate(4-6); 4,Severe(7-10) 10.

In case of moderate to severe postoperative pain, the patients were instructed to take a capsule of placebo given to him/her at the end of each visit. In case of persistent pain, patients were allowed to take Ibuprofen 400mg. The incidence of placebo intake and number of analgesic tablets taken were recorded by the patients.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults of 18-50 years. The diagnosis of symptomatic irreversible pulpitis with symptomatic apical periodontitis in a posterior mandibular tooth was confirmed by history of chief complaint of moderate to severe lingering sharp throbbing pain with pain on biting, clinical examination revealing positive response to an electrical pulp tester and tenderness to percussion on tapping the tooth with the end of a mirror handle, and radiographic examination showing posterior tooth with no apical radiolucency or slight widening of lamina dura.

Exclusion Criteria:

* pregnant women, patients who reported bruxism or clenching, or patients who have administrated analgesics preoperatively during the past 12 hours that might alter their pain perception. Teeth that had no occlusal contact, no sensitivity to percussion, association with swelling or fistulous tract, greater than grade I mobility, or no possible restorability were also excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
postinstrumentation pain | up to 48 hours following instrumentation
  postoperative pain was measured using visual analogue scale (VAS) following root canal instrumentation
postobturation pain | upto 24 hours following obturation
  postoperative pain was measured using visual analogue scale (VAS) following root canal obturation

SECONDARY OUTCOMES:
incidence of placebo and analgesic intake | up to 48 hours following each visit
  The incidence of placebo intake and number of analgesic tablets taken were recorded by the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Radwa S Emara, Masters, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No
IPD data are confidential and secured. Only accessed by principal investigator and supervisors